CLINICAL TRIAL: NCT02713035
Title: Behavioral Self-Help Intervention for Pediatric Atopic Dermatitis and Eczema Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: moved to new institution
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Stephanie jacks, Assistant Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0172
Record Dates: First submitted 2016-03-09; First posted 2016-03-18 (Estimated); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Dermatitis, Atopic; Eczema
MeSH Terms: conditions — Dermatitis, Atopic; Eczema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual (No Intervention): Receive standard medical therapy for eczema
- Treatment (Experimental): Receive standard medical therapy for eczema plus behavioral self help intervention
  Interventions: Behavioral: Self help intervention

INTERVENTIONS:
Behavioral: Self help intervention — For participants randomized to receive the treatment, the self-help intervention will be briefly described by a member of the clinical staff, and a brief pamphlet will be distributed to the parent or guardian at the end of the visit. The pamphlet describes behavioral strategies for coping with and reducing scratching behaviors. Participants randomly selected to not receive the treatment will not receive the pamphlet at the end of the visit.
  Arms: Treatment

SUMMARY:
Patients with atopic dermatitis and eczema often struggle with habitual scratching that is not well-controlled even with optimal medical therapy. Our goal is to create a behavioral intervention to help children with eczema reduce scratching. The investigators hope that the intervention will improve clinical outcomes and quality of life, as well as provide an easily implemented way for clinicians to educate patients and parents about behavioral modification techniques.

DETAILED DESCRIPTION:
Background Psychological interventions for atopic dermatitis (AD) in children are not well-studied, despite the potential benefits, which may include: decreased need for medications and improved long-term control of both dermatologic symptoms as well as other secondary symptoms that may impact quality of life, such as anxiety, insomnia, and psychosocial distress. Chida and colleagues (2007) conducted a meta-analysis of psychological interventions for AD. Of the eight studies that were included in the meta-analysis, only four studies examined pediatric patients. A wide-range of psychological interventions were evaluated, including cognitive-behavioral therapy, stress management programs, aromatherapy massage, psychodynamic therapy, and structured educational programs focusing on a wide range of medical and psychological topics (e.g., nutrition, relaxation). Seven of the eight studies showed some positive effects on measures of eczema severity, scratching/itching, use of topical steroids, and anxiety.

More recently, Ersser and colleagues (2014) evaluated the literature on psychological and educational interventions for AD focusing on studies conducted among children. Ten randomized controlled trials were reviewed, including 9 educational interventions and one study that evaluated a psychological intervention.Particular promise in terms of modest improvement in disease severity and quality of life was noted in a large study (N=992) that utilized a multidisciplinary group education intervention in an inpatient setting. However, the authors of the review concluded that there is a lack of research on this topic. Accordingly, additional studies evaluating psychological and educational interventions are needed. Previous studies have evaluated time- and resource-intensive interventions that may not be practical outside of a randomized controlled trial or a large academic research setting. Nevertheless, adjunctive psychological interventions are promising for reducing symptoms associated with severe dermatologic issues. To address this gap, the current study will evaluate the utility and acceptability of a brief self-help behavioral intervention in a pilot study, which emphasizes the effectiveness of the study design. A brief self-help intervention that utilizes well-supported cognitive and behavioral psychological strategies will be distributed to interested patients and families to augment the standard skin-directed treatments for eczema or AD. The self-help intervention will be distributed to and discussed with a family in less than five minutes in an outpatient clinic setting by clinical staff with no special training in psychology. The target population is children with AD aged 4-12 years with prominent excoriations and their guardians. At the standard 1-4 month follow-up visit, feasibility and acceptability of the self-help intervention will be assessed. Brief evaluations of medical and behavioral symptoms will be conducted at the initial visit and the follow-up.

Purpose The purpose of the current study is to pilot a brief self-help behavioral intervention that will be implemented in conjunction with treatment as usual in children with AD or eczema between the ages of 4 and 12 years. The acceptability and effectiveness of the intervention will be evaluated. The intervention aims to reduce the severity of AD or eczema symptoms and improve the quality of life in children. It is hypothesized that the adjunctive self-help behavioral treatment will reduce the severity of eczema and improve quality of life for patients who receive the intervention compared to patients who only receive standard dermatologic treatment. Additionally, itching intensity, scratching behaviors, and anxiety symptoms will be included as outcome measures.

Specific Aims Aim 1: Pilot a brief self-help behavioral intervention to be delivered to children with eczema or AD and their parents.

Aim 2: Evaluate feasibility and acceptability of a brief self-help behavioral intervention.

Aim 3: Evaluate effectiveness of the self-help intervention for reducing symptom severity and improving quality of life.

Study Period This study will occur over a two year period from July 1, 2015 thru June 30, 2017. Interested patients will receive the treatment information at the first appointment and then a follow up visit will be conducted 1-4 months later.

Study Methodology Study Design This will be a randomized, case-controlled, prospective trial that compares treatment as usual to treatment as usual with the addition of the brief self-help intervention. Half of the patients will receive the self-help intervention and the other half will not receive the self-help intervention. A priori block randomization procedures will be conducted in attempt to secure an equal distribution of participants in each condition. The block randomization involves randomizing blocks of 6-8 participant numbers, where half of the participants in the treatment as usual group and half of the participants in the treatment group. Then, the order of the blocks are randomized. The physician (Dr. Jacks) recruiting participants will be blind to the condition until after the patient has consented to participate. All patients will receive the standard of care for eczema or atopic dermatitis, which may include dry skin care with emollients, topical steroids, topical calcineurin inhibitors, and oral antihistamines. All patients will undergo initial evaluation and then a follow up evaluation at 1-4 months later.

Research Participants (N = 150) Children between the ages of 4 and 12 and their parents who are presenting to the UMMC pediatric dermatology clinic will be invited to participate in the study. It is anticipated that 75 parent-child dyads will enroll in the study procedures, for a total of 75 children and 75 parents.

Inclusion criteria Inclusion criteria: (1) children presenting to the pediatric dermatology clinic; (2) current or new diagnosis of eczema or AD; (3) between the ages of 4 and 12; and (4) excoriation is reported by the patient or parent or noted by the clinical staff to be a prominent issues within the past month.

Exclusion criteria Exclusion criteria: (1) inability to complete English-language questionnaires; (2) patients requiring systemic immunosuppressives such as systemic prednisone, methotrexate, azathioprine, mycophenolate mofetil, or cyclosporine; (3) Patients with known comorbidities that cause immunodeficiency, such as HIV, treatment with chemotherapy, or genetic syndromes; (4) Patients who are being treated by a mental health provider (e.g., counselor, psychologist) or psychiatrist for issues specifically related to excoriation.

Procedure. Recruitment will occur through the UMMC pediatric dermatology clinic. Clinical staff will identify potential study participants through Epic database searches and chart reviews of eczema and atopic dermatitis pediatric patients seen in the UMMC Dermatology Clinic practice. The treating physician (Dr. Jacks) will approach potential participants either by phone or in person at the clinic to inform them of the study and its procedures and to see if they are interested in participating. If interested, screening criteria will be reviewed with the patients and their parents. If the patient is eligible for the study, they will be invited to participate in the study. Consent, parent permission, and child assent will be obtained children and their parents.

At the initial visit, after the patient has received standard care or while in the examination room waiting for standard care, the patients and their parents will complete several brief self-report questionnaires that will take approximately 10 minutes to complete. These questionnaires will assess socio-demographic information, symptom intensity, quality of life, anxiety symptoms, and symptom severity. A priori randomization will determine whether the participant receives the self-help intervention or not. For participants randomized to receive the treatment, the self-help intervention will be briefly described by a member of the clinical staff, and a brief pamphlet will be distributed to the parent or guardian at the end of the visit. The pamphlet describes behavioral strategies for coping with and reducing scratching behaviors. Participants randomly selected to not receive the treatment will not receive the pamphlet at the end of the visit. A routine follow-up appointment will be scheduled with all patients, which is typically scheduled 1-4 months after the initial visit. This is a routine follow-up interval for children with active eczema or AD.

At the follow-up visit, verbal consent for the follow up assessment will be obtained from participants. Patients and their parents who provide verbal consent will complete a second set of brief self-report questionnaires in the waiting room or while in the examination room. The questionnaires are expected to take approximately 10 minutes to complete. The questionnaires will include measures assessing acceptability and feasibility of the self-help intervention, quality of life, anxiety symptoms, and dermatology symptom severity (i.e., SCORAD). For patients who are unable to come in for the follow-up visit, typical clinical procedures for following up with a missed appointment will be followed. Additional attempts to contact the participant will be made by the research personnel to contact the parents by telephone to either to complete the questionnaires over the telephone or to come in for the brief follow up study visit. If participants chose to attend the study session, but not the follow up dermatology appointment, then they would not receive the standard care visit, but would only complete the study procedures and accordingly would not be billed. If the participant expresses that they are not interested in participating in the follow up study visit, study personnel will cease attempts at study contact and follow up.

Measures. Screener. A brief screener will be conducted with the patient and the parent to verify eligibility in the study per the inclusion and exclusion criteria.

Assessment of Co-variates Socio-demographics Form. The parents/guardians of patients will be asked questions related to their and their child's demographics, including age, race, marital status, socioeconomic status, and medical history (including current medications).

ELIGIBILITY:
Inclusion Criteria:

1. children presenting to the pediatric dermatology clinic;
2. current or new diagnosis of eczema or AD;
3. between the ages of 4 and 12;
4. excoriation is reported by the patient or parent or noted by the clinical staff to be a prominent issues within the past month.

Exclusion Criteria:

1. inability to complete English-language questionnaires;
2. patients requiring systemic immunosuppressives such as systemic prednisone, methotrexate, azathioprine, mycophenolate mofetil, or cyclosporine;
3. Patients with known comorbidities that cause immunodeficiency, such as HIV, treatment with chemotherapy, or genetic syndromes;
4. Patients who are being treated by a mental health provider (e.g., counselor, psychologist) or psychiatrist for issues specifically related to excoriation.

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
SCORAD - Scoring Atopic Dermatitis - change at follow-up 1-4 months later | Baseline and Follow up visit - change at follow-up 1-4 months later
  widely-used, validated tool for quantifying the extent and severity of eczema. The form is completed by the physician evaluating the patient in the office, and we will plan to complete this measure at both the initial and follow-up visit.
Index of Itching Intensity and Scratching Activity - change at follow-up 1-4 months later | Baseline and Follow up visit - change at follow-up 1-4 months later
  5-item self-report questionnaire that assesses current and past week intensity of itching, frequency of scratching behaviors, and excoriations occurring as a result of scratching. This measure will be completed at both the initial and follow-up visit.
Acceptability and Feasibility Questionnaire- to assess at follow-up 1-4 months later | the follow-up visit in 1-4 months to participants who received the self-help intervention
  The 11-item questionnaire obtains self-report feedback from the parent with regard to: acceptability of the pamphlet, ease of readability, and use of the pamphlet.

SECONDARY OUTCOMES:
Children's Dermatology Quality of Life Index | Baseline and Follow up visit - change at follow-up 1-4 months later
  well-validated measure comprised of 10 items measuring health-related quality of life over the previous week among pediatric dermatology patients
Preschool Anxiety Scale - Parent Report (PAS) or the Spence Children's Anxiety Scale-Parent Report (SCAS) - depending on patient age | Baseline and Follow up visit- change at follow-up 1-4 months later
  The PAS and the SCAS are well-validated, self-report measures that are commonly utilized for the clinical assessment of anxiety symptoms in children. The PAS-Parent Version is validated to assess symptoms among children between 3 and 5 years, and the SCAS is utilized for children between 6 and 18 years. The measures are not diagnostic instruments, but indicate the severity of a range of anxiety symptoms. The PAS is completed by a parent and includes 34 items that assess anxiety symptoms on a 0 (not true at all) to 4 (Very often true) scale. Similarly, the SCAS-Parent Version is a 39-item scale measuring child anxiety on six different domains. The items are rated by the parent on a likert scale from 0 (Never) to 3 (Always). Total and subscale scores are computed by adding the corresponding items.
Child Anxiety Sensitivity Index - Parent Version | Baseline and Follow up visit- change at follow-up 1-4 months later
  18-item measure that assesses fear of anxiety symptoms in children per parent report. Anxiety sensitivity is a well-supported transdiagnostic factor that contributes to mental health and health conditions in children and adults. Items are rated by the parent on a three-point scale (0 = none; 1 = some; 2 = a lot). An example question is "It scares my child when she/he feels nervous." The total score is computed by adding the items

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie K Jacks, MD, Principal Investigator — assistant professor
Locations (1):
- Pavilion Dermatology Suite K, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No
All data will be reviewed by a member of the research team the same week it is collected in order to ensure completion and clarity. The research team will maintain an updated data tracking form indicating when participant data are collected, entered, and verified, as well as any corrections that are needed. The PI, clinical staff, and trained bachelors- or Master-level staff will collect the data, and will thus have access to participant identities. However, the investigators will safeguard against breaches of confidentiality by coding participant data by ID number rather than by name, and by keeping information linking these ID numbers to specific individuals in a locked file cabinet accessible only to project staff. Further, individuals will not be identified by name (nor will any identifying information be offered) when results from data are disseminated.